CLINICAL TRIAL: NCT05019898
Title: Comparison Between Pupillometry and the Numerical Rating Scale for the Assessment of Pain in Communicating Adult Patients Presenting to the Emergency Room.
Brief Title: Comparison Between Pupillometry and the Numerical Rating Scale
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEWC_MAYS2021
Record Dates: First submitted 2021-08-10; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pain, Acute
Keywords: pupillometry
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Test: pupillometry (Experimental)
  Interventions: Diagnostic Test: pupillometry

INTERVENTIONS:
Diagnostic Test: pupillometry — Step 1: The triage will be carried out by the nurse. The nurse will then perform a self-assessment of the patient's pain using a simple verbal scale.
  The nurse will then record the patient's self-assessment of his pain using the numeric scale for pain.
  Step 2: Immediately after this first assessment, eligible patients will be approached by the study investigator to be included in the study.
  Step 3: If the patient gives informed consent, the study investigator will perform
  * The quantification of their anxiety
  * An assessment of pain by a NeuroLight videopupillometer (iDmed, Marseille, France) using two dynamic tests, the Pupillary Unrest in Ambient Light (PUAL) and the pupillary light reflex.
  Step 4: One hour after the triage, a second pain assessment will be performed. Step 5: The same pupillometry measurements will be taken immediately after the nurse has assessed the pain.

SUMMARY:
Given the difficulties encountered with subjective pain assessment tools, one of the ideas for reducing the occurrence of insufficient analgesia administration in the emergency department is to find a tool capable of measuring pain without requiring the patient's participation, and which could be integrated into the systematic measurement of the 4 other vitals. An interesting idea is the measurement of pupillary diameter and its reflex variations by a portable pupillometer. Indeed, the diameter of the pupil (DP) reflects the constant interactions between the sympathetic and parasympathetic systems at the level of the iris muscles. Pupillometry measures the change in pupillary diameter and allows the performance of three dynamic tests useful in the assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the emergency room, aged 18 years or over, able to communicate, with hemodynamic and respiratory stability, are eligible.

Exclusion Criteria:

* - Refusal to participate in the study; refusal to sign informed consent.
* Consent impossible to obtain (cognitive disorders, language barrier…).
* Patient taking immediate-release opioid medication (last dose within the last 12 hours).
* Patient taking prolonged-release opioid medication (last dose within the last 24 hours).
* Basic treatment with a dopaminergic D2 antagonist (antipsychotic drugs).
* Basic treatment with dopamine antagonist antiemetic medication (metoclopramide (T1/2 5-6h), domperidone (T1/2 7-9h), alizapride (T1/2 3h)) within the last 12 hours.
* Patient taking clonidine (last dose within the last 24 hours).
* Use of topical ocular drugs modifying pupillary parameters in the last 24 hours.
* Bilateral eye surgery modifying the possibilities of variation in pupillary diameter bilaterally.
* Parkinson's or Alzheimer's disease at a dysautonomic stage.
* Admission to the emergency room for acute ocular pathology.
* History of diabetes at a dysautonomic stage.
* History of alcoholism at a dysautonomic stage.
* History of glaucoma.
* Pregnant patient with preeclampsia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the correlation between the pupillometry values and those obtained by the numerical pain rating scale with a correlation coefficient of 0.78. | 1 minute

SECONDARY OUTCOMES:
The evolution of the Pupillary Unrest in Ambient Light depending on the type of opioid (morphine versus weak opioid like tramadol) received by the patient. | one hour
The endpoint will be the evaluation of the performance of pupillometry to predict the occurrence of Numerical Rating Scale (NRS) ≥ 4 using the ROC curve (AUC). | 1 minute
The correlation of the pupillometric parameters with the level of anxiety quantified by a numeric scale next to 1 (not anxious) to 10 (maximum level of anxiety). | 1 minute
The correlation between the initial measurement of PUAL and the analgesic response to an opioid medication. | one hour
The correlation between the pain measurements obtained by the reception nurse and that obtained by the patient. | 2 minutes
The evolution of the pupillary light reflex depending on the type of opioid (morphine versus weak opioid like tramadol) received by the patient. | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregoire C, Charier D, de Bergeyck R, Mouraux A, Van Ouytsel F, Lambert R, Zhou N, Lavand'homme P, Penaloza A, Pickering G. Comparison between pupillometry and numeric pain rating scale for pain assessments in communicating adult patients in the emergency department. Eur J Pain. 2023 Sep;27(8):952-960. doi: 10.1002/ejp.2137. Epub 2023 Jun 11. PMID 37303073